CLINICAL TRIAL: NCT06215222
Title: Capsule Microbiota Sampling in IBS/Functional Gastrointestinal Disease
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Spencer, Instructor, Stanford University
Other Study IDs: IRB-62670
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: IBS - Irritable Bowel Syndrome; Healthy; Functional Bloating; Functional Gastrointestinal Disorders
Keywords: microbiome; Small intestine
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy patients: Healthy Patients
  Interventions: Other: Microbiota Sampling
- IBS/Functional GI diasease: Patients with IBS or Functional GI disease (bloating, diarrhea, constipation)
  Interventions: Other: Microbiota Sampling

INTERVENTIONS:
Other: Microbiota Sampling — We will sample the Saliva, Feces, and intestinal microbiome for genetic microbiome analysis and bacterial isolation

SUMMARY:
We will sample intestinal microbiota using a microbiome sampling capsule in Healthy, Irritable Bowel Syndrome (IBS), and Functional Gastrointestinal Disease.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 years of age or older and 70 years of age or younger at the time of the first Screening Visit.
* American Society of Anesthesiologists (ASA) Physical Status Classification System 1 or 2 (1-A normal healthy patient or 2-A patient with mild systemic disease)
* For women of childbearing potential, negative urine pregnancy test within 7 days of Screening Visit. Willingness to use highly effective contraception during the entire study period (e.g.: implants, injectables, oral contraceptives, intra-uterine device or declared abstinence).
* Subject is fluent in English and understands the study protocol and informed consent and is willing and able to comply with study requirements and sign the informed consent form.
* Positive for at least one clinical symptoms consistent with SIBO and or IBS and or a Rome Diagnosis of functional GI disorder (Rome IV criteria)

Exclusion Criteria:

* History of any of the following:

  * Prior gastric or esophageal surgery, including lap banding or bariatric surgery
  * Bowel obstruction
  * Gastric outlet obstruction
  * Diverticulitis
  * Inflammatory bowel disease
  * Ileostomy or colostomy
  * Gastric or esophageal cancer
  * Achalasia
  * Esophageal diverticulum
* Active Dysphagia or Odynophagia
* Active medication use for any gastrointestinal conditions
* Pregnancy or planned pregnancy within 30 days from Screening Visit, or breast-feeding
* Any form of active substance abuse or dependence (including drug or alcohol abuse), unstable medical or psychiatric disorder, or any chronic condition susceptible, in the opinion of the investigator, to interfere with the conduct of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Subjects or those with clinical symptoms consistent with SIBO and or IBS and or a Rome Diagnosis of functional GI disorder (Rome IV criteria)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Collection of 50ul of intestinal fluid from >90% of microbiome sampling capsules | 1-4 years
  Collection of 50ul of intestinal fluid from microbiome sampling capsules

SECONDARY OUTCOMES:
Isolation of liven bacteria from the intestinal fluid of >90% of microbiome sampling capsules | 1-4 years
  Isolation of liven bacteria from the intestinal fluid of >90% of microbiome sampling capsules

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Digestive Health Clinic, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: Undecided